CLINICAL TRIAL: NCT05345379
Title: A Clinical Comparison of the Effectiveness of Two Moisture Insensitive Primers on Orthodontic Attachment Bond: A Randomized Clinical Trial
Brief Title: A Clinical Comparison of the Effectiveness of Two Moisture Insensitive Primers on Orthodontic Attachment Bond
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ahmed Abdulelah Abduljawad, orthodontics master student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 594422
Record Dates: First submitted 2022-04-13; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Dental Bonding
Keywords: moisture insensitive primers; orthodontic; molar tube; bond failure rate; Assure plus bond; Transbond MIP
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: The primers will be randomly allocated using a split-mouth, cross-quadrant design. In each patient, two diagonal quadrants (i.e. upper right and lower left, or vice versa) will be randomly assigned to each primer group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial will be triple-blinded in which neither the participants nor the trial team will know which one of the primers a patient has received, as well as the outcome assessor will be blinded. This can be achieved by placing the two primers in two similar masked bottles and giving them numerical coding i.e. number one and number two coding for either type of primer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transbond MIP (Experimental): Transbond primer group will be randomly allocated using a split-mouth, cross-quadrant design and two diagonal quadrants (i.e. upper right and lower left, or vice versa) for each participant.
  Interventions: Other: Single intervention
- Assure plus (Experimental): Assure Plus primer group will be randomly allocated using a split-mouth, cross-quadrant design and two diagonal quadrants (i.e. upper right and lower left, or vice versa) for each participant.
  Interventions: Other: Single intervention

INTERVENTIONS:
Other: Single intervention — Single intervention at the day of fixed orthodontic appliance bonding

SUMMARY:
A single-operator, randomized controlled trial (RCT) will be conducted to evaluate the clinical effectiveness of moisture insensitive primers (MIPs) in bonding molar tubes under moisture contaminated conditions by comparing the clinical bond failure and survival rate of molar tubes using two MIPs which are Transbond ™ MIP (3M Unitek Dental Products, Monrovia, CA, USA) and Assure® Plus-All Surface Light Cure Bonding Primer (Reliance, Itasca, IL, USA).

DETAILED DESCRIPTION:
A single-operator, a multi-centre, a split-mouth, cross-quadrant RCT, with 1:1 allocation ratio will be conducted for patients seeking for orthodontic treatment with fixed orthodontic appliance. The study will be conducted at postgraduate Orthodontic Clinic/ College of Dentistry/University of Baghdad in addition to private dental clinics in Baghdad, Iraq. Patients seeking for orthodontic treatment and their treatment will be planned with metal fixed orthodontic appliance (0.22" for both arches) will be recruited for this trial. Patients who will met the eligible criteria will be randomly assigned to either group of primer type. A single operator to avoid inter-operator variation will bond all molar tubes. A standardized protocol of tooth preparation and molar tubes bonding will be adopted for all the patients. All teeth will be isolated and cleansed with a mixture of water and pumice using a rubber-polishing cup on a low speed hand piece. The teeth will be rinsed and dried with an oil-free air syringe, and will be etched with the conventional acid etching technique (37% orthophosphoric acid applied for 30sec). They will be subsequently rinsed thoroughly with water for 10sec to ensure total removal of etchant according to the manufacturer's instructions.

Without drying, one coat of the patient own non-stimulated saliva will be applied to the etched and wet surface using bond brush; the excess will be blotted with a moist cotton pellet maintaining the surface moist.

A liberal coat of the MIP will be applied to the etched area of the teeth destined for a specific primer (split-mouth) using a nylon bond brush. Air will be gently blown on each tooth for 2sec, aiming the air stream perpendicular to the enamel surface then light cured for 20sec. After etching and priming, molar tubes will be bonded to the teeth with a light-cured adhesive according to the manufacturer's instructions.

Initial wires will be fitted 10-15mins after bonding completion in the context of the straight wire technique.

All patients will receive the same instructions and will be seen at 3-4-week intervals. They will be, however, requested to inform the operator immediately and attend as soon as possible once a bond failure was apparent. the molar tubes bond survival will be followed up for 6 months. They will be instructed to brush with a manual toothbrush using a fluoride-containing toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking for metal fixed orthodontic appliance with 0.22"*0.28";
* Complete set of permanent dentition with fully erupted molar teeth on both arches;
* Intact 1st molars and mainly their buccal surfaces are free from caries, fillings, or gingival hyperplasia;

Exclusion Criteria:

* Patients with systemic problem or genetic syndrome that affecting enamel surface like patients with generalized enamel hypoplasia.
* Patients exhibit parafunctional habits;
* Patients who their treatment plan need appliance that soldered on molar bands.
* No occlusal interferences that can affect the ideal position of molar tubes, especially in the lower arch.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Clinical bond failure rate | First 6 months
  the number of times in which bond failure of molar tubes happens over a period of time (6 months).

SECONDARY OUTCOMES:
Adhesive remnant index (ARI) | First 6 months
  determines the amount of adhesive remaining on the tooth surface when bond failure occurs.
Bond failure location in the dental arch. | First 6 months
  correlations between upper and lower arches and right and left sides with bond failure rate

OTHER OUTCOMES:
Age | First 6 months
  correlations of age with bond failure rate
Gender | First 6 months
  correlations of gender with bond failure rate

CONTACTS AND LOCATIONS:
Overall Officials: Harraa S Abdulameer, B.D.S, PhD, Study Director — Baghdad college of dentistry, Department of orthodontics; Ahmed A Abduljawad, B.D.S, Principal Investigator — Baghdad college of dentistry, Department of orthodontics
Locations (1):
- Baghdad college of dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD because this trial is a prospective study and yet we can't promise for any sharing.

REFERENCES:
- [Background] Zeppieri IL, Chung CH, Mante FK. Effect of saliva on shear bond strength of an orthodontic adhesive used with moisture-insensitive and self-etching primers. Am J Orthod Dentofacial Orthop. 2003 Oct;124(4):414-9. doi: 10.1016/s0889-5406(03)00405-0. PMID 14560272
- [Background] Endo T, Ozoe R, Sanpei S, Shinkai K, Katoh Y, Shimooka S. Effects of moisture conditions of dental enamel surface on bond strength of brackets bonded with moisture-insensitive primer adhesive system. Odontology. 2008 Jul;96(1):50-4. doi: 10.1007/s10266-007-0083-7. Epub 2008 Jul 27. PMID 18661205
- [Background] Goswami A, Mitali B, Roy B. Shear bond strength comparison of moisture-insensitive primer and self-etching primer. J Orthod Sci. 2014 Jul;3(3):89-93. doi: 10.4103/2278-0203.137695. PMID 25143933
- [Background] Paschos E, Westphal JO, Ilie N, Huth KC, Hickel R, Rudzki-Janson I. Artificial saliva contamination effects on bond strength of self-etching primers. Angle Orthod. 2008 Jul;78(4):716-21. doi: 10.2319/0003-3219(2008)078[0716:ASCEOB]2.0.CO;2. PMID 18302473
- [Background] Roelofs T, Merkens N, Roelofs J, Bronkhorst E, Breuning H. A retrospective survey of the causes of bracket- and tube-bonding failures. Angle Orthod. 2017 Jan;87(1):111-117. doi: 10.2319/021616-136.1. Epub 2016 Jun 15. PMID 27304230
- [Background] Hadrous R, Bouserhal J, Osman E. Evaluation of shear bond strength of orthodontic molar tubes bonded using hydrophilic primers: An in vitro study. Int Orthod. 2019 Sep;17(3):461-468. doi: 10.1016/j.ortho.2019.06.006. Epub 2019 Jul 2. PMID 31278045
- [Background] Gange P. The evolution of bonding in orthodontics. Am J Orthod Dentofacial Orthop. 2015 Apr;147(4 Suppl):S56-63. doi: 10.1016/j.ajodo.2015.01.011. PMID 25836345
- See also: Transbond MIP product page — https://3m.com/3M/en_US/p/d/b5005137018/
- See also: Assure plus product page — https://www.relianceorthodontics.com/Assure-Plus

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT05345379/Prot_SAP_ICF_000.pdf